CLINICAL TRIAL: NCT01628809
Title: Stress Reduction and Healthy Living in Pittsburgh
Brief Title: Mindfulness-Based Meditation to Treat Stress in Unemployed Community Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, David Creswell, Dr. J. David Creswell, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLS-2011
Record Dates: First submitted 2012-06-20; First posted 2012-06-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Stress; Inflammation
Keywords: MBSR; mindfulness; stress
MeSH Terms: conditions — Inflammation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rest and Relaxation (Active Comparator): three-day relaxation retreat without mindfulness components
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Mindfulness-Based Meditation (Experimental): three-day mindfulness-based meditation retreat
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — three-day mindfulness-based meditation retreat program
  Other Names: MBSR

SUMMARY:
The purpose of this study is to determine the effects of a three-day mindfulness meditation retreat (vs. a three-day relaxation retreat) in stressed, unemployed, community adults on brain function, brain structure, and overall health and immunity.

DETAILED DESCRIPTION:
Chronic stress has been shown to be a significant risk factor for increased morbidity and mortality. Eight-week Mindfulness-Based Meditation programs (MBSR) have been shown to improve participants' health and well-being, including reducing inflammation and slowing the progression of chronic diseases such as HIV. The purpose of this study is to evaluate the potential benefits of a three-day mindfulness-based meditation retreat program (vs. an active rest and relaxation retreat control condition) on a highly stressed, unemployed, community adult population.

Participants are recruited from the Pittsburgh area and are randomly assigned to either the mindfulness-based retreat program or the rest and relaxation retreat program. All participants complete a psychosocial survey, blood work, and a baseline fMRI before completing the intervention. Participants complete a second fMRI immediately following the intervention and then additional blood work and psychosocial surveys at a four month follow-up timepoint. At each fMRI appointment, participants will complete neuroimaging tasks (where they will be presented with words, picture, and sounds) that will assess neuroreactivity, regulation responses, and brain volume before and after mindfulness meditation training.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults between the ages of 24 and 52 years at time of entry
* non-pregnant women only
* currently unemployed
* high levels of self-reported stress
* geographically accessible and willing to travel to and attend all study sessions

Exclusion Criteria:

* not able to attend scheduled three-day retreat
* have regularly (>1 time per week) practiced a mind-body therapy anytime in the last six months (e.g., meditation, yoga, tai chi)
* indicate any major physical health problems in the last six months
* have more than 15 alcoholic drinks in the average week
* have been diagnosed with a chronic disease (e.g. HIV, diabetes, arthritis)
* use medications affecting cardiovascular or endocrine function
* are left-handed
* have metal in their bodies (including pacemakers and permanent piercings (e.g., bellyrings, but not dental fillings))
* indicate regular use of psychotropic medication or psychotherapy in the last six months
* cognitive impairment as indicated by a score lower than 23 on the Mini-Mental State examination
* demonstrate low levels of stress due to unemployment
* smokers
* indicate use of recreational drugs in the past month
* indicate feeling claustrophobic in confined spaces, such as an fMRI scanner
* weigh over 350 lbs
* have any neurological disorders
* indicate any use of doctor prescribed cholesterol lowering medications (e.g., statins)
* currently employed
* not currently looking for a job

Ages: 24 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Functional Neural Activity | Change from randomization to 1 week
  Neural response to emotionally evocative stimuli including stressors related to be unemployed

SECONDARY OUTCOMES:
Brain volume | Change from randomization to 1 week
  Change in volume of brain areas associated with emotional reactivity
Pro-inflammation | from baseline to four-month follow-up
  Change in protein measures of inflammation
Psychological Distress | baseline to four month follow-up
  self-reported psychological distress
Cortisol Levels | 1 day
  Levels of cortisol were assessed from a small sample of participants' hair

CONTACTS AND LOCATIONS:
Overall Officials: J. David Creswell, PhD, Principal Investigator — Carnegie Mellon University

REFERENCES:
- [Derived] Taren AA, Gianaros PJ, Greco CM, Lindsay EK, Fairgrieve A, Brown KW, Rosen RK, Ferris JL, Julson E, Marsland AL, Creswell JD. Mindfulness Meditation Training and Executive Control Network Resting State Functional Connectivity: A Randomized Controlled Trial. Psychosom Med. 2017 Jul/Aug;79(6):674-683. doi: 10.1097/PSY.0000000000000466. PMID 28323668
- [Derived] Creswell JD, Taren AA, Lindsay EK, Greco CM, Gianaros PJ, Fairgrieve A, Marsland AL, Brown KW, Way BM, Rosen RK, Ferris JL. Alterations in Resting-State Functional Connectivity Link Mindfulness Meditation With Reduced Interleukin-6: A Randomized Controlled Trial. Biol Psychiatry. 2016 Jul 1;80(1):53-61. doi: 10.1016/j.biopsych.2016.01.008. Epub 2016 Jan 29. PMID 27021514
- [Derived] Taren AA, Gianaros PJ, Greco CM, Lindsay EK, Fairgrieve A, Brown KW, Rosen RK, Ferris JL, Julson E, Marsland AL, Bursley JK, Ramsburg J, Creswell JD. Mindfulness meditation training alters stress-related amygdala resting state functional connectivity: a randomized controlled trial. Soc Cogn Affect Neurosci. 2015 Dec;10(12):1758-68. doi: 10.1093/scan/nsv066. Epub 2015 Jun 5. PMID 26048176